CLINICAL TRIAL: NCT03657043
Title: Open Label Phase 2 Study of Tisotumab Vedotin for Patients With Platinum-Resistant Ovarian Cancer With a Safety Run-in of a Dose-Dense Regimen
Brief Title: A Study of Weekly Tisotumab Vedotin for Patients With Platinum-Resistant Ovarian Cancer With Safety Run-in (innovaTV 208)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNTV-002
Record Dates: First submitted 2018-08-22; First posted 2018-09-04 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Platinum-resistant; Antibody drug conjugate; Tisotumab vedotin; PROC; Seattle Genetics
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — tisotumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Run-In (3Q4W Schedule) (Experimental): 28-day, 3 dose cycle
  Interventions: Drug: tisotumab vedotin
- Part A: Tisotumab Vedotin (Experimental): 21-day, single dose cycle
  Interventions: Drug: tisotumab vedotin
- Part A: Tisotumab Vedotin (3Q4W Schedule) (Experimental): 28-day, 3 dose cycle
  Interventions: Drug: tisotumab vedotin
- Part B: Tisotumab Vedotin (3Q4W Schedule) (Experimental): 28-day, 3 dose cycle
  Interventions: Drug: tisotumab vedotin

INTERVENTIONS:
Drug: tisotumab vedotin — Intravenous (IV) infusion
  Other Names: TIVDAK

SUMMARY:
This trial will study tisotumab vedotin to find out what its side effects are and to see if it works for platinum-resistant ovarian cancer (PROC). It will test different doses of tisotumab vedotin that are given at different times. It will also compare the side effects and ability to treat tumors of these different doses and schedules. In this study, there will be a safety run-in group of approximately 12 patients that will look at a dose-dense treatment schedule. In a dose-dense schedule, smaller doses are given more frequently. In addition to the safety run-in patients, there will be three groups in the study. One group will get tisotumab vedotin once every 3 weeks (21-day cycles). The two other groups will get tisotumab vedotin once a week for 3 weeks followed by 1 week off (28-day cycles).

DETAILED DESCRIPTION:
The study objectives are to evaluate the safety, antitumor activity, and pharmacokinetics of tisotumab vedotin (TV) administered every 3 weeks or on Days 1, 8, and 15 of every 4-week cycle (3Q4W) for patients with epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer that has relapsed within 6 months of the completion of platinum-based treatment and determined to be platinum resistant. All patients must have PROC and be eligible for single agent chemotherapy.

The safety run-in period will evaluate the safety of a weekly schedule. The highest dose level that is considered safe will be the recommended phase 2 dose (RP2D) and will be used in Part A. In Part A, participants will be randomized in a 1:1 ratio to receive tisotumab vedotin intravenously (IV) every 3 weeks (Q3W regimen) or the safety run-in RP2D on Days 1, 8, and 15 of every 4-week cycle (weekly regimen; 3Q4W) if a RP2D has been identified. Participants who enroll in Part B will receive tisotumab vedotin on Days 1, 8, and 15 of every 4-week cycle (weekly regimen) at a pre-specified dose level, if the dose level is considered safe and tolerable in the safety run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
* Safety run-in only: PROC. Patients may have received more than 1 prior systemic treatment regimen in the PROC setting.
* Part A and Part B only: Patients with PROC who have received 1 to 3 anticancer lines of therapy overall, including at least 1 line of therapy containing bevacizumab or biosimilar.

  * Adjuvant ± neoadjuvant are considered 1 line of therapy.
  * Patients may have received a PARP inhibitor or an immuno-oncology (IO) agent; any of these regimens are to be considered a line of therapy for the purposes of this study if not used as maintenance therapy.
  * Maintenance therapy (including bevacizumab, PARP inhibitors and IOs) will be considered part of the preceding line of therapy and not to be counted as a new line of therapy.
  * Any chemotherapy regimen change due to toxicity in the absence of disease progression is considered as part of the same line of therapy.
  * Hormonal therapy will be not be counted towards the lines of therapy.
* Measurable disease according to RECIST v1.1 as assessed by the investigator
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1
* Life expectancy of at least 3 months
* Able to provide fresh or archival tissue for biomarker analysis

Exclusion Criteria:

* Primary platinum-refractory disease, defined as disease progression within 2 months of completion of first line platinum-based therapy
* Patients with clinical symptoms or signs of gastrointestinal obstruction with the past 6 months or who currently require parenteral nutrition
* Hematological: Known past or current coagulation defects leading to an increased risk of bleeding, diffuse alveolar hemorrhage from vasculitis, known bleeding diathesis, ongoing major bleeding, or trauma with increased risk of life-threatening bleeding within 8 weeks of trial entry
* Cardiovascular: Clinically significant cardiac disease including uncontrolled hypertension, unstable angina, acute myocardial infarction with 6 months of screening, serious cardiac arrhythmia requiring medication, medical history of congestive heart failure, or medical history of decreased cardiac ejection fraction of <45%
* Ophthalmological: Active ocular surface disease at baseline or prior episode of cicatricial conjunctivitis or Stevens Johnson syndrome
* Prior treatment with MMAE-derived drugs
* Inflammatory bowel disease including Crohn's disease and ulcerative colitis
* Ongoing, acute, or chronic inflammatory skin disease
* Uncontrolled tumor-related pain
* Inflammatory lung disease requiring chronic medical therapy
* Grade 3 or higher pulmonary disease unrelated to underlying malignancy
* Uncontrolled pleural or pericardial effusions
* Grade >1 peripheral neuropathy
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Schmidt, MD, Study Director — Seagen Inc.
Locations (37):
- United States (21):
  - Stanford Cancer Center South Bay, San Jose, California
  - Poudre Valley Health System (PVHS), Fort Collins, Colorado
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Miami Cancer Institute- Plantation (MCIP), Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - University of Missouri Healthcare / Ellis Fischel Cancer Center, Columbia, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, The, Cleveland, Ohio
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - Cleveland Clinic Hillcrest Hospital, Mayfield Heights, Ohio
  - Texas Oncology - Fort Worth, Dallas, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - University of Virginia, Charlottesville, Virginia
- Belgium (2):
  - Algemeen Ziekenhuis Maria Middelares, Ghent, Other
  - Universitair Ziekenhuis Leuven, Lueven, Other
- Aalborg Universite Hospital, Aalborg, Other, Denmark
- Ireland (2):
  - Mater Private, Dublin, Other
  - Cork University Hospital, Wilton, Other
- Italy (5):
  - Ospedale Ramazzini di Carpi, Carpi, Other
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori- IRST S.r.l, Meldola, Other
  - Istituto Europeo di Oncologia, Milan, Other
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Other
  - Fondazione Policlinico Universitario Agostino, Rome, Other
- Spain (6):
  - Hospital Universitario Vall d'Hebron, Barcelona, Other
  - L'Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Other
  - Hospital Universitario Ramon y Cajal, Madrid, Other
  - HM Centro Integral Oncologico Clara Campal, Madrid, Other
  - Clinica Universidad de Navarra, Pamplona, Other
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Other

REFERENCES:
- [Derived] Feng S, Gunawan R, Passey C, Voellinger J, Polhamus D, Gerritsen A, O'Day C, Carret AS, Soumaoro I, Gupta M, Hanley WD. Exposure-safety Markov modeling of ocular adverse events in patient populations treated with tisotumab vedotin. J Pharmacokinet Pharmacodyn. 2025 Oct 3;52(5):55. doi: 10.1007/s10928-025-10003-w. PMID 41044356

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 98 participants were enrolled into the Safety Run-In and Part B Expansion cohorts, of which 94 received study drug. No participants were enrolled into Part A.
Groups:
- Safety Run-In 0.9 mg/kg 3Q4W; Part B Expansion: Tisotumab Vedotin 0.9 mg/kg by IV infusion on Days 1, 8, and 15 of every 4-week cycle
- Safety Run-In 1.2 mg/kg 3Q4W: Tisotumab Vedotin 1.2 mg/kg by IV infusion on Days 1, 8, and 15 of every 4-week cycle
- Part A Q3W: Tisotumab Vedotin 2.0 mg/kg by IV infusion on Day 1 of each 3-week treatment cycle
- Part A 3Q4W: Tisotumab Vedotin by IV infusion on Days 1, 8, and 15 of every 4-week cycle
Period: Overall Study
Arm/Group | Safety Run-In 0.9 mg/kg 3Q4W | Safety Run-In 1.2 mg/kg 3Q4W | Part A Q3W | Part A 3Q4W | Part B Expansion
Started | 8 | 8 | 0 | 0 | 82
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 8 | 8 | 0 | 0 | 82
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 4
Not completed — Study closure by Sponsor | 0 | 2 | 0 | 0 | 17
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 4
Not completed — Death | 6 | 5 | 0 | 0 | 53
Not completed — Met exclusion criteria after enrollment | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal - subsequent treatment | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal - declined follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set includes all participants who received any amount of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run-In 0.9 mg/kg 3Q4W | Safety Run-In 1.2 mg/kg 3Q4W | Part B Expansion | Total
Number analyzed (Participants) | 7 | 8 | 79 | 94
Age, Continuous [Median (Full Range); unit: Years] | 69.0 [50.0 to 87.0] | 67.5 [51.0 to 74.0] | 60.0 [38.0 to 81.0] | 62.0 [38.0 to 87.0]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 7 | 8 | 79 | 94
  Intersex | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 6 | 7
  White | 6 | 6 | 69 | 81
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino/a, or of Spanish Origin | 0 | 1 | 9 | 10
  Not of Hispanic or Latino/a, or of Spanish Origin | 6 | 7 | 69 | 82
  Unknown | 1 | 0 | 1 | 2
Eastern Cooperative Oncology Group (ECOG) Performance Score [Count of Participants; unit: Participants] — Measure Description: 0=Normal activity; 1=Symtoms but ambulatory; 2=In bed <50% of the time; 3= In bed > 50% of the time; 4=100% bedridden; 5=Dead
  Participants
    Grade 0 | 4 | 5 | 48 | 57
    Grade 1 | 3 | 3 | 31 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) (Safety Run-In Only)
Description: Incidence of dose-limiting toxicity (DLT) was evaluated in participants enrolled in the Safety Run-In, who were followed for protocol-defined DLT events up to 28 days after the first dose of tisotumab vedotin.
Time Frame: Up to 28 days
Population: Participants from the Safety Analysis Set that were enrolled in the Safety Run-In. The Safety Analysis Set includes all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In 0.9 mg/kg 3Q4W | Safety Run-In 1.2 mg/kg 3Q4W
Number analyzed (Participants) | 7 | 8
Participants | 0 | 1

2. Primary Outcome: Confirmed Objective Response Rate (ORR) (Part B)
Description: Proportion of participants who achieve a confirmed complete response (CR) or partial response (PR) according to RECIST v1.1 as assessed by the investigator
Time Frame: Up to 9.7 months
Population: The Full Analysis Set includes all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Expansion
Number analyzed (Participants) | 79
Participants | 7

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) (Part B)
Description: An AE is any untoward medical occurrence in a patient or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Treatment emergent AEs (TEAEs) are defined as events that are new or worsened on or after receiving the first dose of study treatment and up through 30 days after the last dose of study treatment.
Time Frame: Up to 23.0 months
Population: The Safety Analysis Set includes all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Expansion
Number analyzed (Participants) | 79
Participants
  Any TEAE | 79
  Treatment-related TEAE | 67
  Treatment-related Grade 3-4 TEAE | 14
  Treatment-related Grade 5 TEAE | 0
  Max severity of TEAE - Grade 1 | 7
  Max severity of TEAE - Grade 2 | 35
  Max severity of TEAE - Grade 3 | 32
  Max severity of TEAE - Grade 4 | 3
  Max severity of TEAE - Grade 5 | 2
  Any treatment-emergent serious AE (SAE) | 28
  Treatment-related SAE | 6

4. Secondary Outcome: Confirmed and Unconfirmed ORR (Part B)
Description: Proportion of participants who achieve a CR or PR according to RECIST v1.1 as assessed by the investigator
Time Frame: Up to 9.7 months
Population: The Full Analysis Set includes all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B Expansion
Number analyzed (Participants) | 79
Percentage of Participants | 18.0 [10.0 to 27.9]

5. Secondary Outcome: Cancer Antigen 125 (CA-125) Response Rate According to Gynecologic Cancer Intergroup (GCIG) Criteria (Part B)
Description: Percentage of participants who have at least a 50% reduction in CA-125 value from baseline
Time Frame: Up to 10.1 months
Population: The CA-125 evaluable analysis set includes participants who have an elevated baseline CA-125 value of ≥2 x ULN (upper limit of normal) within 2 weeks prior to the first dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B Expansion
Number analyzed (Participants) | 51
Percentage of Participants | 12.0 [4.4 to 23.9]

6. Secondary Outcome: Overall Response According to the Gynecological Cancer Intergroup (GCIG) Combined RECIST and CA-125 Criteria (Part B)
Description: Percentage of participants whose best response is a CR or PR according to the GCIG combined RECIST and CA-125 criteria
Time Frame: Up to 10.1 months
Population: The Full Analysis Set includes all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B Expansion
Number analyzed (Participants) | 79
Percentage of Participants | 11.0 [5.3 to 20.5]

7. Secondary Outcome: Duration of Response (DOR) (Part B)
Description: Time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the first documentation of PD or death due to any cause, whichever comes first
Time Frame: Up to 8.3 months
Population: Subset of the Full Analysis Set includes all participants who received any amount of study drug and had a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B Expansion
Number analyzed (Participants) | 7
Months | 4.21 [3.02 to NA] — Upper limit not available, insufficient number of events.

8. Secondary Outcome: Disease Control Rate (DCR) (Part B)
Description: Percentage of participants who achieved a confirmed Complete Response(CR) or Partial Response (PR) per RECIST v1.1 as assessed by the investigator, or meet the Stable Disease (SD) criteria at least once after start of study treatment at a minimum interval of 12 weeks.
Time Frame: Up to 3.0 months
Population: The Full Analysis Set includes all participants who received any amount of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part B Expansion
Number analyzed (Participants) | 79
Percentage of Participants | 54.4 [42.8 to 65.7]

9. Secondary Outcome: Time to Response (TTR) (Part B)
Description: Time from the start of study treatment to the first documentation of objective response (CR or PR that is subsequently confirmed)
Time Frame: Up to 23.0 months
Population: as for outcome 7
Measure: Median (Full Range); unit: Months
Arm/Group | Part B Expansion
Number analyzed (Participants) | 7
Months | 1.4 [1.0 to 3.0]

10. Secondary Outcome: Progression-free Survival (PFS) (Part B)
Description: Time from the start of study treatment to the first documentation of PD or death due to any cause, whichever comes first
Time Frame: Up to 9.7 months
Population: The Full Analysis Set includes all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B Expansion
Number analyzed (Participants) | 79
Months | 2.73 [1.64 to 2.99]

11. Secondary Outcome: Overall Survival (OS) (Part B)
Description: Time from the start of study treatment to date of death due to any cause
Time Frame: Up to 23.0 months
Population: The Full Analysis Set includes all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part B Expansion
Number analyzed (Participants) | 79
Months | 10.68 [7.75 to 12.81]

12. Secondary Outcome: Incidence of Antitherapeutic Antibodies (ATA) (Part B)
Description: The proportion of participants who develop ATA at any time during the study. A positive baseline ATA result is considered positive post-baseline if the post-baseline ATA titer result is at least four times higher than the baseline result.
Time Frame: Up to 6.9 months
Population: Participants in the Safety Analysis Set with a baseline and at least one post-baseline ATA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Expansion
Number analyzed (Participants) | 71
Participants
  Baseline Negative - Negative post-baseline | 65
  Baseline Negative - Positive post-baseline | 3
  Baseline Positive - Negative post-baseline | 3
  Baseline Positive - Positive post-baseline | 0

13. Secondary Outcome: Pharmacokinetic (PK) Parameter: Antibody-Drug Conjugate (ADC) Maximum Concentration (Cmax) (Part B)
Description: ADC Cmax was derived from the PK blood samples collected.
Time Frame: Samples for PK measures were collected at Cycle 1 Day 1 (predose, end of infusion, 1 hr, and 5 hr), Day 3, Day 8 (predose), Day 15 (predose, end of infusion, 1 hr, and 5 hr), Day 17, Day 22, and Cycle 2 Day 1 (predose). Approximately 4 weeks per cycle.
Population: PK analysis set which includes enrolled participants who received any amount of study drug and at least one PK parameter can be estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
µg/mL
  Cycle 1, Dose 1 | 20.582 (26.963)
  Cycle 1, Dose 3 | 21.817 (26.823)

14. Secondary Outcome: PK Parameter: ADC Time of Cmax (Tmax) (Part B)
Description: ADC Tmax was derived from the PK blood samples collected.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
Days
  Cycle 1, Dose 1 | 0.041 (53.112)
  Cycle 1, Dose 3 | 0.041 (78.407)

15. Secondary Outcome: PK Parameter: ADC Area Under Concentration-Time Curve (AUC) (Part B)
Description: ADC AUC was derived from the PK blood samples collected.
Time Frame: Cycle 1 Dose 1 AUC 7: Assessed from Cycle 1 Days 1 - 8 (predose). Cycle 1 Dose 3 AUC 7: Assessed from Cycle 1 Days 15 - 22. Cycle 1 Dose 3 AUC 14: Assessed from Cycle 1 Days 15 - Cycle 2 Day 1 (predose).
Population: PK Analysis Set includes enrolled participants who received any amount of study drug and at least one PK parameter can be estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL*day
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
µg/mL*day
  Cycle 1, Dose 1 - AUC 7 Days-ADC | 25.198 (25.335)
  Cycle 1, Dose 3 - AUC 7 Days-ADC | 30.159 (32.261)
  Cycle 1, Dose 3 - AUC 14 Days-ADC | 31.716 (31.632)

16. Secondary Outcome: PK Parameter: Free Monomethyl Auristatin E (MMAE) Cmax (Part B)
Description: MMAE Cmax was derived from the PK blood samples collected.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
ng/mL
  Cycle 1, Dose 1 | 1.778 (66.636)
  Cycle 1, Dose 3 | 2.552 (52.442)

17. Secondary Outcome: PK Parameter: MMAE Tmax (Part B)
Description: MMAE Tmax was derived from the PK blood samples collected.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
Days
  Cycle 1, Dose 1 | 2.061 (26.838)
  Cycle 1, Dose 3 | 2.101 (28.820)

18. Secondary Outcome: PK Parameter: MMAE AUC (Part B)
Description: MMAE AUC was derived from the PK blood samples collected.
Time Frame: as for outcome 13
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*day
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
ng/mL*day
  Cycle 1, Dose 1 - AUC Last-MMAE | 8.709 (63.747)
  Cycle 1, Dose 3 - AUC Last-MMAE | 16.578 (52.121)

19. Secondary Outcome: PK Parameter: MMAE Trough Concentration (Ctrough) (Part B)
Description: MMAE Ctrough was derived from the PK blood samples collected.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
ng/mL | 0.230 (82.638)

20. Secondary Outcome: PK Parameter: Total Antibody (TAb) Cmax (Part B)
Description: TAb Cmax was derived from the PK blood samples collected.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
ng/mL
  Cycle 1, Dose 1 | 18.418 (28.631)
  Cycle 1, Dose 3 | 19.955 (28.405)

21. Secondary Outcome: PK Parameter: TAb Tmax (Part B)
Description: TAb Tmax was derived from the PK blood samples collected.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
Days
  Cycle 1, Dose 1 | 0.041 (67.072)
  Cycle 1, Dose 3 | 0.043 (67.795)

22. Secondary Outcome: PK Parameter: TAb Area Under Concentration-Time Curve (AUC) (Part B)
Description: TAb AUC was derived from the PK blood samples collected.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL*day
Arm/Group | Part B Expansion
Number analyzed (Participants) | 77
µg/mL*day
  Cycle 1, Dose 1 - AUC 7 Days-TAb | 35.535 (24.950)
  Cycle 1, Dose 3 - AUC 7 Days-TAb | 39.371 (29.218)
  Cycle 1, Dose 3 - AUC 14 Days-TAb | 42.240 (29.206)

ADVERSE EVENTS:
Time Frame: Non-serious AEs were followed up to 10.5 months. Serious AEs and All-Cause Mortality were followed up to 31.6 months.
Description: All-cause mortality includes all participants that were enrolled in the study regardless of whether or not they received treatment. Non-serious AEs and SAEs were collected and reported for patients that received treatment in their respective arms.
Arm/Group | Safety Run-In 0.9 mg/kg 3Q4W | Safety Run-In 1.2 mg/kg 3Q4W | Part B Expansion
All-Cause Mortality (participants affected / at risk) | 6/8 | 5/8 | 53/82
Serious Adverse Events (participants affected / at risk) | 2/7 | 4/8 | 28/79
Other Adverse Events (participants affected / at risk) | 7/7 | 8/8 | 77/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In 0.9 mg/kg 3Q4W (N=7) | Safety Run-In 1.2 mg/kg 3Q4W (N=8) | Part B Expansion (N=79)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In 0.9 mg/kg 3Q4W (N=7) | Safety Run-In 1.2 mg/kg 3Q4W (N=8) | Part B Expansion (N=79)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 0 (0) | 23 (33)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 7 (9)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctival ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 12 (14)
Ectropion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Entropion (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 5 (8)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 4 (9)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 7 (8)
Punctate keratitis (Eye disorders) | 0 (0) | 2 (2) | 2 (2)
Symblepharon (Eye disorders) | 0 (0) | 1 (1) | 4 (4)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 9 (10)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 8 (9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 22 (27)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 1 (1) | 6 (7)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (4) | 17 (20)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 18 (25)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 30 (37)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1) | 15 (19)
Asthenia (General disorders) | 0 (0) | 0 (0) | 19 (23)
Fatigue (General disorders) | 2 (2) | 4 (4) | 25 (27)
Malaise (General disorders) | 0 (0) | 1 (2) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 5 (5)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 6 (16)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (3) | 1 (1) | 25 (33)
Conjunctivitis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pustule (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 5 (6)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 5 (5)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1)
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 6 (6)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 5 (7)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 25 (29)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 8 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 14 (17)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 10 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 7 (7)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (5)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 5 (5)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 2 (3) | 18 (20)
Restless legs syndrome (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (6)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 5 (6)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 6 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 9 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 36 (46)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 9 (9)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 10 (10)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT03657043/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03657043/SAP_001.pdf